CLINICAL TRIAL: NCT04531553
Title: The Impact of Ultrasound-Guided Erector Spinae Plane Block Versus Thoracic Epidural Analgesia in the Management of Acute and Chronic Post-Thoracotomy Pain: A Randomized, Controlled Study
Brief Title: Erector Spinae Plane Block for Post-thoracotomy Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Assistant professor of Anesthesia, intensive care and pain releif, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESPB for PTPS
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Post-thoracotomy Pain Syndrome
MeSH Terms: interventions — Tea; Levobupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic epidural analgesia (Active Comparator): Patients will preoperatively receive thoracic epidural at the level T5 & T6 with bolus 20 ml of levobupivacaine 0.25% then levobupivacaine 0.1% infused at a rate of 0.1 mL/Kg/h until chest tube removal ( 5-6 days).
  Interventions: Procedure: Thoracic epidural analgesia
- ESPB with levobupivacaine (Active Comparator): patients will preoperatively receive US guided ESP block on the side to be operates upon, the puncture point of the skin is infiltrated with 2% lidocaine, and once the structures are identified with ultrasound at the level of T5 transverse process, we will inject bolus 20ml of levobupivacaine 0.25% on the deep aspect of erector spinae muscle then catheter inserted.A 20 ml bolus of levobupivacaine 0.1% is injected every 6 hours until chest tube removal.
  Interventions: Procedure: ESPB with levobupivacaine
- ESPB with levobupivacaine and dexmedetomidine (Active Comparator): patients will preoperatively receive US guided ESP block on the side to be operates upon, the puncture point of the skin is infiltrated with 2% lidocaine, and once the structures are identified with ultrasound at the level of T5 transverse process, we will inject bolus 20ml of levobupivacaine 0.25% plus 0.5mic/Kg dexmedetomidine on the deep aspect of erector spinae muscle then catheter inserted. 20 ml bolus of levobupivacaine 0.1% with dexmedetomidine 0.5 μg/Kg was injected every 6 hours until chest tube removal.
  Interventions: Procedure: ESPB with levobupivacaine and dexmedetomedine

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — Patients will preoperatively receive thoracic epidural at the level T5 & T6 with bolus 20 ml of levobupivacaine 0.25% then levobupivacaine 0.1% infused at a rate of 0.1 mL/Kg/hr until chest tube removal ( 5-6 days).
  Arms: Thoracic epidural analgesia
Procedure: ESPB with levobupivacaine and dexmedetomedine — patients will preoperatively receive US guided ESP block on the side to be operates upon, the puncture point of the skin is infiltrated with 2% lidocaine, and once the structures are identified with ultrasound at the level of T5 transverse process, we will inject bolus 20ml of levobupivacaine 0.25% plus 0.5mic/Kg dexmedetomidine on the deep aspect of erector spinae muscle then catheter inserted. 20 ml bolus of levobupivacaine 0.1% with dexmedetomidine 0.5 μg/Kg was injected every 6 hours until chest tube removal.
  Arms: ESPB with levobupivacaine and dexmedetomidine
Procedure: ESPB with levobupivacaine — patients will preoperatively receive US guided ESP block on the side to be operates upon, the puncture point of the skin is infiltrated with 2% lidocaine, and once the structures are identified with ultrasound at the level of T5 transverse process, we will inject bolus 20ml of levobupivacaine 0.25% on the deep aspect of erector spinae muscle then catheter inserted.A 20 ml bolus of levobupivacaine 0.1% is injected every 6 hours until chest tube removal.
  Arms: ESPB with levobupivacaine

SUMMARY:
The thoracic epidural block (TEB) and thoracic paravertebral block (TPVB) are the most commonly used techniques for analgesia after thoracic surgery.Recently, erector spinae plane block (ESPB) was reported as a treatment for thoracic neuropathic pain.Dexmedetomidine has been primarily used for intra- venous sedation in intensive care settings. The unique analgesic properties of dexmedetomidine have encouraged the anesthesiologists to use it perineurally.

This study aims to evaluate the effect ultrasound erector spinae plane block with dexmedetomidine infusion in management of acute and chronic post thoracotomy pain.

DETAILED DESCRIPTION:
The thoracic epidural block (TEB) and thoracic paravertebral block (TPVB) are the most commonly used techniques for analgesia after thoracic surgery. However, TEA has several adverse effects, such as hypotension, motor blockade, hematoma, and abscess and TPVB has a chance of epidural spread and pneumothorax, and multiple injections are needed if more than 4 dermatome analgesia is required. Recently, erector spinae plane block (ESPB) was reported as a treatment for thoracic neuropathic pain.

ESPB is a relatively simple technique with easily identified sonographic landmarks, and a catheter is easily inserted into the plane after distention induced by the injection. Additionally, the ESPB has the potential to provide both somatic and visceral sensory blockade.

The selectivity of dexmedetomidine to the α2-receptors is eight times of its prototype, clonidine. Accordingly, dexmedetomidine is a more powerful sedative and analgesic drug than clonidine with less hemodynamic derangements from the α1-receptor activation. Dexmedetomidine has been primarily used for intra- venous sedation in intensive care settings. The unique analgesic properties of dexmedetomidine have encouraged the anesthesiologists to use it perineurally. Previous studies have declared that dexmedetomidine potentiates local anesthetic effect when administered by neuroaxial route.

This study aims to evaluate the effect ultrasound erector spinae plane block with dexmedetomidine infusion in management of acute and chronic post thoracotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA I and II.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.
* Patient undergoing thoracotomy for cancer surgery (Lobectomy, Pneumonectomy, and Decortication).

Exclusion Criteria:

* Patient refusal
* Known sensitivity or contraindication to local anesthetics or dexmedetomidine.
* History of psychological disorders.
* Localized infection at the site of block.
* Coagulopathies with platelet count below 50,000 or an INR>1.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity score | 1 week
  measurement of Visual analogue score in a line 0 to 100 , where 0 indicates no pain and 100 indicates the worst pain.

SECONDARY OUTCOMES:
Number of patients who will develop post-thoracotomy pain syndrome. | 3 months
  Reporting the emergence of post-thoracotomy pain syndrome in all the studied patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Gendy, MD, Principal Investigator — Assistant Professor of Anesthesia, intensive care and pain releif
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
After submitting the paper authors are planning to share IPD